CLINICAL TRIAL: NCT02718547
Title: The Effect of Reducing the Intraocular Pressure by Using Alphagan Drops and Macular Edema in Patients With Diabetic Macular Edema
Brief Title: The Relationship Between Intraocular Pressure and Macular Edema in Patients With Diabetic Macular Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Meir Hospital, Kfar Saba, Israel (Other)
Responsible Party: Principal Investigator, Avner Belkin, MD, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0029-16-MMC
Record Dates: First submitted 2016-03-06; First posted 2016-03-24 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Complications of Diabetes Mellitus
Keywords: Diabetes mellitus; Diabetic macular edema; Intra ocular pressure; Ocular perfusion pressure; Retinal perfusion
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination; Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving Combigan drops in order to reduce IOP (Experimental): All of the Participants in this study will be instructed to instill combigan eye drops twice daily in one eye (randomly chosen)
  Interventions: Drug: Combigan

INTERVENTIONS:
Drug: Combigan — Each Participant will be instructed to instill Combigan eye drops twice daily in one of his eyes (randomly chosen)
  Other Names: brimonidine tartrate/timolol maleate ophthalmic solution

SUMMARY:
The Investigators propose to examine the effect of lowering the intraocular pressure on macular edema in Participants diagnosed with diabetic macular edema. Our theory is based on the assumption that lower intraocular pressure means higher Ocular Perfusion pressure, which may cause an improvement in retinal perfusion and thus an improvement in retinal oxygenation and reduced edema

DETAILED DESCRIPTION:
Ocular perfusion pressure (ocular perfusion pressure - OPP), considered the driving force of ocular blood flow. Perfusion pressure is defined as the difference between the artery and vein blood pressure. Because ocular venous pressure is the same or slightly higher than the IOP (intra ocular pressure - IOP), it is common to estimate the OPP as the difference between the arterial blood pressure of IOP. The OPP is critical for diffusion of oxygen, nutrients and metabolic waste from retinal imaging, and decrease it may reduce blood flow to the eye and lead to ischemia or hypoxia. the OPP is controlled by a complex system of Autoregulation. Much has been written about the relationship between the OPP and glaucoma, and agreed that OPP is a low risk factor for this disease.

Diabetic macular edema (DME) is the most common cause of vision loss in developed countries the working-age.

Many studies were carried out in recent years in an attempt to better understand the pathophysiology of Diabetic macular edema, and there is consensus in the scientific literature that hypertension have a significant effect on Diabetic macular edema. this relationship is much more complex than it seems at first glance. Paques and his team have shown an inverse association between blood pressure to drop night and Diabetic macular edema. LARSEN and his team have shown a similar trend.

Hayreh published an article from 2007, where he described the mechanism of improvement of the Diabetic macular edema with discontinuation of hypertensive treatment and thereby raising blood pressure. In this article, Hayreh describes hypoxia as a significant factor in Diabetic macular edema, and demonstrated that treatment of hypoxia by increasing the OPP brought good results in terms of macular thickness If so, it seems that there is not only a link between levels of oxygenation of the retina to Diabetic macular edema, but that improved oxygenation of the retina could lower the levels of macular edema in these patients. If a way were found to improve retinal perfusion, this may lead to an improved oxygenation and reduced edema. The Investigators propose to examine the relationship between macular edema IOP in Participants with Diabetic macular edema, thinking that high IOP means lower OPP, which means increased risk for developing macular edema in this Participants group.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of diabetic macular edema over the age of 18 which are eligible to sign an agreement to participate in the study
* Presence of DME (based on clinical examination of retinal specialist + OCT) in both eyes with an edema thickness ranged from 350 to 800 microns
* Media lucid enough to allow sufficient quality photographs by OCT

Exclusion Criteria:

* Patients which do not have a valid diagnosis of DME (Diabetic Macular Edema)
* Patients with problems that can cause macular edema in any other:

  * Age-Related Macular Degeneration
  * Central retinal vein occlusion (CRVO)/Branch retinal vein occlusion (BRVO) /central retinal artery occlusion (CRAO) / branch retinal artery occlusion (BRAO)
  * Epiretinal membrane (ERM) or Vitreo-macular traction (VMT)
  * Patients who are Pseudophakic in one eye or pseudophakic in both eyes for less than a year
  * Patients treated in order to reduce the DME by intra-vitreal injection or by laser in the past six months
  * Patients which are currently treat with Intra ocular Pressure lowering drops in at least one eye, or have been treated in the past with laser of any kind or with surgery
  * Patients who underwent Pars plana vitrectomy one or both eyes
  * Patients who cannot undergo an OCT examination
  * Patients who want prefer to be treated by the current practices based on clinical judgment
  * Patients with a condition that requires an intervention or laser surgery during the 3 months of study, such as active Proliferative diabetic retinopathy, vitreous hemorrhage or other similar conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-03-26 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change of at least 50 micron in Macular edema | Baseline measurement will be conducted at the recruitment of the participant, the second measurement will be preformed after one moth from recruitment and the third and last measurement will be preformed after 3 months from recruitment
  The participants will be examined every month from the time of recruitment as mentioned before, at each visit the Macular Edema will be assessed, but the Outcome measure will be defined as Change of at least 50 Micron in Macular Edema at the third visit, 3 months from recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical center, Kfar Saba, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glucksberg MR, Dunn R. Direct measurement of retinal microvascular pressures in the live, anesthetized cat. Microvasc Res. 1993 Mar;45(2):158-65. doi: 10.1006/mvre.1993.1015. PMID 8361399
- [Background] Schmidl D, Garhofer G, Schmetterer L. The complex interaction between ocular perfusion pressure and ocular blood flow - relevance for glaucoma. Exp Eye Res. 2011 Aug;93(2):141-55. doi: 10.1016/j.exer.2010.09.002. Epub 2010 Sep 22. PMID 20868686
- [Background] Thomas BJ, Shienbaum G, Boyer DS, Flynn HW Jr. Evolving strategies in the management of diabetic macular edema: clinical trials and current management. Can J Ophthalmol. 2013 Feb;48(1):22-30. doi: 10.1016/j.jcjo.2012.11.012. PMID 23419295
- [Background] Lasker RD. The diabetes control and complications trial. Implications for policy and practice. N Engl J Med. 1993 Sep 30;329(14):1035-6. doi: 10.1056/NEJM199309303291410. No abstract available. PMID 8366905
- [Background] Klein R, Klein BE, Moss SE, Cruickshanks KJ. The Wisconsin Epidemiologic Study of Diabetic Retinopathy. XV. The long-term incidence of macular edema. Ophthalmology. 1995 Jan;102(1):7-16. doi: 10.1016/s0161-6420(95)31052-4. PMID 7831044
- [Background] Bhagat N, Grigorian RA, Tutela A, Zarbin MA. Diabetic macular edema: pathogenesis and treatment. Surv Ophthalmol. 2009 Jan-Feb;54(1):1-32. doi: 10.1016/j.survophthal.2008.10.001. PMID 19171208
- [Background] Matthews DR, Stratton IM, Aldington SJ, Holman RR, Kohner EM; UK Prospective Diabetes Study Group. Risks of progression of retinopathy and vision loss related to tight blood pressure control in type 2 diabetes mellitus: UKPDS 69. Arch Ophthalmol. 2004 Nov;122(11):1631-40. doi: 10.1001/archopht.122.11.1631. PMID 15534123
- [Background] Paques M, Massin P, Sahel JA, Gaudric A, Bergmann JF, Azancot S, Levy BI, Vicaut E. Circadian fluctuations of macular edema in patients with morning vision blurring: correlation with arterial pressure and effect of light deprivation. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4707-11. doi: 10.1167/iovs.05-0638. PMID 16303968
- [Background] Larsen M, Wang M, Sander B. Overnight thickness variation in diabetic macular edema. Invest Ophthalmol Vis Sci. 2005 Jul;46(7):2313-6. doi: 10.1167/iovs.04-0893. PMID 15980216
- [Background] Hayreh SS. Role of retinal hypoxia in diabetic macular edema: a new concept. Graefes Arch Clin Exp Ophthalmol. 2008 Mar;246(3):353-61. doi: 10.1007/s00417-007-0678-2. Epub 2007 Sep 18. PMID 17876597
- [Background] Vinten M, La Cour M, Lund-Andersen H, Larsen M. Acute effect of pure oxygen breathing on diabetic macular edema. Eur J Ophthalmol. 2012 Aug 8:0. doi: 10.5301/ejo.5000195. Online ahead of print. PMID 22890599
- [Background] Nguyen QD, Shah SM, Van Anden E, Sung JU, Vitale S, Campochiaro PA. Supplemental oxygen improves diabetic macular edema: a pilot study. Invest Ophthalmol Vis Sci. 2004 Feb;45(2):617-24. doi: 10.1167/iovs.03-0557. PMID 14744906
- [Background] Vinten M, la Cour M, Lund-Andersen H, Larsen M. Effect of acute postural variation on diabetic macular oedema. Acta Ophthalmol. 2010 Mar;88(2):174-80. doi: 10.1111/j.1755-3768.2008.01421.x. Epub 2009 Dec 13. PMID 19094166
- [Background] Frederiksen CA, Jeppesen P, Knudsen ST, Poulsen PL, Mogensen CE, Bek T. The blood pressure-induced diameter response of retinal arterioles decreases with increasing diabetic maculopathy. Graefes Arch Clin Exp Ophthalmol. 2006 Oct;244(10):1255-61. doi: 10.1007/s00417-006-0262-1. Epub 2006 Mar 15. PMID 16538448